CLINICAL TRIAL: NCT06316349
Title: Isolated Resistance Training Program Versus Combined With Neuromuscular Electrical Stimulation for Femoral Quadriceps in Patients With Femoral Intra Aortic Balloon Pump: a Randomized Controlled Trial
Brief Title: Isolated Resistance Training and Neuromuscular Electrical Stimulation in Patients With Femoral Intra Aortic Balloon Pump.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rafael M. Ianotti, PT, Clinical Research Coordinator - Physiotherapy Division - Heart Institute (InCor), University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 75727323.3.0000.0068
Record Dates: First submitted 2024-02-19; First posted 2024-03-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Physical Therapy; Neuromuscular Electrical Stimulation
Keywords: Heart Failure; Intra-Aortic Ballom Pump; Acquired Muscle Weakness; Neuromuscular Electrical Stimulation; Muscular echo intensity
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Rondomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The researcher responsible for conducting the ultrasonographic measurements will be blinded regarding the randomization and allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated Resistance Training Program Group (Active Comparator): Four sets of 10 knee extension repetitions will be performed with a 90-second rest interval between sets.
  Interventions: Other: Isolated Resistance Training Program
- Neuromuscular Electrical Stimulation Group (Experimental): Neuromuscular electrical stimulation will be performed in muscles of the femoral quadriceps, simultaneously with the same resistance exercise program as the Isolated Resistance Training Program Group.
  Interventions: Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Isolated Resistance Training Program — The hip range of motion (ROM) will be fixed at 45 degrees due to the limitation imposed by the femoral insertion of the intra-aortic balloon pump in both lower limbs to allow for a 45-degree knee extension ROM. Four sets of 10 knee extension repetitions will be performed with a 90-second rest interval between sets. The intensity (resistive load) will be set at 60% of the baseline load, calculated using the one-repetition maximum (1RM) test and increased by 10% after every 5 interventions.
  Arms: Isolated Resistance Training Program Group
Other: Neuromuscular electrical stimulation — For NMES, two electrodes (area of 5 x 9 cm) will be positioned perpendicular to the muscles of the femoral quadriceps. The parameters of NMES will remain fixed throughout the study: pulsed, biphasic current, with a frequency of 35Hz, pulse width of 1000µs, on-time of 7 seconds (with 3 seconds of rise, 1 second of sustainment, and 3 seconds of descent), and off-time switched off. These settings allow the onset of NMES to be synchronous with the start and end of hip extension for simultaneous execution with resistance exercises and a total of 40 stimulations. The intensity will be gradually adjusted until evoked contractions of grade 4 to 5 (partial muscle recruitment and total muscle recruitment) or the maximum intensity tolerated by the patient is achieved.
  Arms: Neuromuscular Electrical Stimulation Group

SUMMARY:
The objective of this randomized clinical trial is to compare the effects of a standardized exercise program alone versus the same program combined with neuromuscular electrical stimulation in patients undergoing heart failure . The main questions it aims to answer are:

* Assessing the ultrasonographic parameters: echo intensity (echogenicity), cross-sectional area, thickness, and pennation angle of the rectus femoris muscle in both lower limbs.
* Evaluating the strength of the femoral quadriceps muscle
* Evaluating the changes in the chronaxie of the rectus femoris muscle in both lower limbs.

The protocol will have a total duration of 32 days, with an initial intervention period of 18 days, followed by a 14-day follow-up period.

DETAILED DESCRIPTION:
- Introduction: Patients with refractory heart failure who develop cardiogenic shock may require the use of an intra aortic balloon pump. This device, when inserted through the femoral artery, necessitates bed rest and increases the incidence of muscle mass loss. Rehabilitation programs in the intensive care unit that include resistive training bring benefits such as improving muscle architecture, strength, and function. Neuromuscular electrical stimulation (NMES) can be an important tool to assess excitability and improve muscle strength through muscle contractions generated by motor axon depolarization. Muscle ultrasonography is currently used as a tool for evaluating and monitoring muscle architecture (echointensity) and mass.

- Objectives: To evaluate the effect of combining NMES with a standardized exercise program on the echointensity (echogenicity) of the rectus femoris muscle in hemodynamically stable patients using an intra aortic balloon pump.

- Method: This is a randomized controlled clinical trial comparing two groups: one group will perform resisted knee extension exercises in both lower limbs, while the other group will perform the same exercises synchronously with NMES of the femoral quadriceps muscle. The resistance load will be determined by the one-repetition maximum test and adjusted if necessary. The intervention period will be 21 days (5 days/week) with a follow-up of 14 days. Muscle architecture and mass (ultrasonography), neuromuscular excitability (using the same NMES device), and knee extension strength (dynamometry) will be assessed at baseline, after 10 and 15 days of intervention and after 14 days from the last intervention day.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Intra-aortic balloon pump (IABP) for more than 48 hours
* Dobutamine ≤ 20 mcg/kg/min
* Norepinephrine ≤ 0.2 mcg/kg/min (35)
* Absence of device failures or bleeding in the last 24 hours
* Mean arterial pressure (MAP) ≥ 60 mmHg and ≤ 120 mmHg
* Heart rate (HR) ≥ 60 bpm and ≤ 120 bpm
* Absence of neurological event with previous cognitive or motor deficit
* Presence of untreated deep venous thrombosis
* Absence of previous autoimmune diseases
* Absence of previous rheumatic diseases

Protocol Discontinuation Criteria:

* Need for norepinephrine > 0.2 mcg/kg/min
* Acute arrhythmia of any etiology with hemodynamic instability
* Hemodynamic instability: MAP < 60 mmHg or >120 mmHg or HR < 60 bpm or > 120 bpm
* Occurrence of neurological event with cognitive or motor deficit

Exclusion Criteria:

* Need for invasive mechanical ventilatory support
* If the patient or responsible family member fails to sign or withdraws the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-03-18 (Estimated); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
To investigate echo intensity of the rectus femoris muscle. | The data will be collected on the day of protocol initiation (baseline), on the first day after the 10th and 15th days of intervention and on the 14th day after the last day of intervention.
  The ultrasonographic images will be obtained by a portable device in B-mode, using a 6 cm linear array transducer with a frequency range of 6-13MHz. The echointensity value will be acquired through quantitative analysis using the square method, in grayscale, where the average value will be calculated using the histogram function of the dedicated software, in arbitrary units (AU).

SECONDARY OUTCOMES:
To investigate cross-sectional area of the rectus femoris muscle. | The data will be collected on the day of protocol initiation (baseline), on the first day after the 10th and 15th days of intervention and on the 14th day after the last day of intervention.
  The cross-sectional area will be determined by the number and size of individual fibers within the rectus femoris muscle, using the measurement of the anatomical area (cross section of a muscle perpendicular to its longitudinal axis) in centimeters square.
To investigate pennation angle of the rectus femoris muscle. | The data will be collected on the day of protocol initiation (baseline), on the first day after the 10th and 15th days of intervention and on the 14th day after the last day of intervention.
  The pennation angle will be calculated by the intersection of the path between the fascia with the lower aponeurosis of the rectus femoris muscle, measured in degrees.
To investigate changes in quadriceps femoral muscle strength. | The data will be collected on the day of protocol initiation (baseline), on the first day after the 10th and 15th days of intervention and on the 14th day after the last day of intervention.
  It will be obtained using digital dynamometry through 3 measurements, with a one-minute interval, and the highest obtained value will be considered, measured in Newtons (N).
To investigate changes in arterial blood pressure during the protocol. | Immediately before and after the end of the protocol.
  Assessed by blood pressure measured by intra aortic baloon pump.
To investigate changes in heart rate during the protocol. | Immediately before and after the end of the protocol.
  Measured by invasive blood pressure monitoring.
To investigate changes in peripheral oxygen saturation during the protocol. | Immediately before and after the end of the protocol.
  Measured by pulse oximetry.
To investigate changes in the veno-arterial difference in carbon dioxide partial pressure. | Immediately before and after the end of the protocol.
  Measured by blood gas analysis sample.
To investigate adverse events: | In each intervention period (5 days a week for 21 days).
  Bleeding at the femoral insertion or changes in the functioning of the IABP, occurrence of acute arrhythmia or hemodynamic instability ( MAP < 60 mmHg or >120 mmHg or HR < 60 bpm or > 120 bpm).

CONTACTS AND LOCATIONS:
Overall Officials: Rafael M Ianotti, PT, Principal Investigator — Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto do Coração - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil